CLINICAL TRIAL: NCT05078580
Title: A Phase 1, Single Dose, Open-label Study to Investigate the Pharmacokinetics and Safety of Iptacopan (LNP023) in Participants With Mild, Moderate, and Severe Hepatic Impairment Compared to Matched Control Healthy Participants With Normal Hepatic Function
Brief Title: Pharmacokinetic (PK) and Safety Study of Iptacopan (LNP023) in Participants With Mild, Moderate, and Severe Hepatic Impairment Compared to Matched Control Healthy Participants With Normal Hepatic Function.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: CLNP023A2105
Record Dates: First submitted 2021-10-13; First posted 2021-10-14 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Hepatic Impairment
Keywords: LNP023; iptacopan; hepatic impairment; single-dose
MeSH Terms: interventions — iptacopan

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healthy participants (Experimental): Iptacopan 200 mg single dose
  Interventions: Drug: Iptacopan
- Mild hepatic impairment patients (Experimental): Iptacopan 200 mg single dose
  Interventions: Drug: Iptacopan
- Moderate hepatic impairment patients (Experimental): Iptacopan 200 mg single dose
  Interventions: Drug: Iptacopan
- Severe hepatic impairment patients (Experimental): Iptacopan 200 mg single dose
  Interventions: Drug: Iptacopan

INTERVENTIONS:
Drug: Iptacopan — Single oral dose of iptacopan 200 mg oral capsules
  Other Names: LNP023
  Arms: Healthy participants
Drug: Iptacopan — Single oral dose of iptacopan 200 mg oral capsules
  Other Names: LNP023
  Arms: Mild hepatic impairment patients
Drug: Iptacopan — Single oral dose of Iptacopan 200 mg oral capsules
  Other Names: LNP023
  Arms: Moderate hepatic impairment patients
Drug: Iptacopan — Single oral dose of Iptacopan 200 mg oral capsules
  Other Names: LNP023
  Arms: Severe hepatic impairment patients

SUMMARY:
This was an open-label, single dose parallel group study to evaluate the PK of iptacopan in participants with mild, moderate, and severe hepatic impairment compared to matched healthy control participants.

DETAILED DESCRIPTION:
The study comprised of a screening period up to 28 days, one Baseline evaluation on Day -1, a single dose administration of 200 mg of iptacopan followed by PK sampling to 240 hr, and an End-of-Study (EOS) visit (Day 11). All participants had a post study safety follow-up call conducted approximately 30 days after last administration of study drug.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this study met the following key criteria:

* Written informed consent was obtained before performing any assessment.
* Male participants and female participants of non-childbearing potential 18 to 75 years of age (inclusive).
* Participants were to weigh at least 55 kg to participate in the study and were to have a body mass index (BMI) within the range of 18 to 35 kg/m2 for healthy participants.

For hepatic impairment participants without overt ascites, the BMI was to be within the range of 18 to 40 kg/m2. For hepatic impairment participants with overt ascites, the BMI was to be within the range of 18 to 45 kg/m2.

* Ability to communicate well with the Investigator, to understand and comply with the requirements of the study.
* Participant was willing to remain in the clinical research unit as required by the protocol

Exclusion Criteria:

Participants meeting any of the following criteria were excluded from this study:

* Use of other investigational drugs within the last 30 days or 5 half-lives prior to dosing, whichever was longer.
* History of hypersensitivity to the investigational compound/compound class or its excipients being used in this study.
* Pregnant or nursing (lactating) women. Pregnancy was defined as the state of a female after conception and until termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test.
* Known history of, or current clinically significant arrhythmias, history of prolonged QT correction formula (QTcF) interval or QTcF > 450 msec (males) or QTcF > 460 msec (females) at screening in healthy participants and history of prolonged QTcF interval or QTcF > 470 msec (males) or QTcF > 480 msec (females) at screening in participants with hepatic impairment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of iptacopan: Cmax The maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration (mass × volume-1) | Day 1 (few time points), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10 and Day 11
  To assess the PK properties of iptacopan after a single oral dose of 200 mg in participants with mild, moderate, or severe hepatic impairment as compared to matched healthy participants with normal hepatic function (Child-Pugh classification).
Pharmacokinetics parameters of iptacopan: Tmax The time to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after single dose administration (time) | Day 1 (few time pints), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10 and Day 11
  To assess the PK properties of iptacopan after a single oral dose of 200 mg in participants with mild, moderate, or severe hepatic impairment as compared to matched healthy participants with normal hepatic function (Child-Pugh classification).
Pharmacokinetic parameters of iptacopan: AUClast The AUC from time zero to the last measurable concentration sampling time (tlast) (mass × time × volume-1) | Day 1 (few time points), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10 and Day 11
  To assess the PK properties of iptacopan after a single oral dose of 200 mg in participants with mild, moderate, or severe hepatic impairment as compared to matched healthy participants with normal hepatic function (Child-Pugh classification).
Pharmacokinetics parameters of iptacopan: AUCinf The AUC from time zero to infinity (mass × time × volume-1) | Day 1 (few time points), Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10 and Day 11
  to assess the PK properties of iptacopan after a single oral dose of 200 mg in participants with mild, moderate, or severe hepatic impairment as compared to matched healthy participants with normal hepatic function (Child-Pugh classification).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Plain Language Trial Summary is available on novctrd.com. — http://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1514